CLINICAL TRIAL: NCT06123949
Title: The Effect of Galvanic Stimulation on vHIT and VEMP Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Berna Özge MUTLU, Principal Inverstigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10840098-604.01.01-41143
Record Dates: First submitted 2023-10-27; First posted 2023-11-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Vestibular System Disorder
Keywords: galvanic vestibular stimulation; VEMP; vHIT
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Galvanic Vestibular Stimulation — Galvanic Vestibular Stimulation (GVS) is a non-invasive technique that uses low-level electrical currents to stimulate the vestibular system, affecting balance, posture, and eye movements. It has applications in research, clinical assessment, and rehabilitation of vestibular and balance-related issues, as well as potential applications in cognitive and motor function enhancement.

SUMMARY:
Introduction: Galvanic vestibular stimulation (GVS) is a well-established technique with a history spanning over a century, primarily used to manipulate the vestibular system. Recent interest has surged in its potential for understanding human vestibular function and aiding in functional recovery. GVS applies electrical currents to the mastoid region, modulating vestibular afferents, and induces specific effects based on the participant's posture and current polarity. While GVS's impact on the central nervous system and its potential to aid in functional recovery have been studied, its immediate effects on vestibular reflexes remain less explored.

Methods: In this study, thirty healthy adult participants underwent ocular and cervical vestibular evoked myogenic potential (VEMP) tests, as well as the velocity Head Impulse Test (vHIT) before and immediately after one hour of GVS application. Statistical analyses were performed to assess changes in VEMP and vHIT results.

ELIGIBILITY:
Inclusion Criteria:

* No history of hearing loss and/or balance disorders
* No physical (neck) problems
* No history of psychological or neurological disorders
* Not using alcohol and/or vestibular suppressant drugs regularly
* Feeling balanced in daily life

Exclusion Criteria:

* History of hearing loss and/or balance disorders
* Physical (neck) problems
* History of psychological or neurological disorders
* Using alcohol and/or vestibular suppressant drugs regularly

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Cervical Vestibuler Evoked Myogenic Potentials | 5 months
  Vestibular evoked myogenic potentials (VEMPs) are muscle reflexes that occur in response to high-intensity acoustic stimuli delivered to the ear. These responses can be easily recorded using surface electrodes placed on the sternocleidomastoid muscle (SCM) or near the inferior oblique muscle .
Ocular Vestibuler Evoked Myogenic Potentials | 5 months
  Vestibular evoked myogenic potentials (VEMPs) are muscle reflexes that occur in response to high-intensity acoustic stimuli delivered to the ear. Ocular VEMP (oVEMP) recorded from surface electrodes placed under the eyes.
Video Head Impulse Test | 5 months
  The vestibulo-ocular reflex (VOR) is responsible for stabilizing images on the fovea during head movement. The velocity Head Impulse Test (vHIT) battery is a standard test for measuring head and eye movements, enabling the calculation of the gain of eye speed. The vHIT system typically employs light goggles to monitor eye position through cameras, along with a gyroscope to measure angular head movements, facilitating the computation of VOR gain.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No